CLINICAL TRIAL: NCT04963335
Title: Effects of a User-centered Exergame Training on Motor and Cognitive Functions in Persons With Multiple Sclerosis: A Pilot Quasi-Randomized Controlled Trial
Brief Title: Effects of a User-centered Exergame Training on Motor and Cognitive Functions in PwMS
Acronym: ExergaMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eling DeBruin (Other)
Responsible Party: Sponsor-Investigator, Eling DeBruin, Prof. Dr., Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BASEC Nr. 2020-02793
Record Dates: First submitted 2021-04-19; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: Exergame; Multiple Sclerosis; Feasibility; Motor functions; Cognitive functions
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants perform 16 exergame training (video game-based physical exercise) sessions over a period of 4 to 8 weeks (depending on in-patient or out-patient). Each training lasts between 15 to 25 minutes. Exergames automatically adjust the game difficulty to the abilities of the respective participant.
  Interventions: Behavioral: Exergame Training
- Control (No Intervention): Participants of the control group are instructed to continue their normal daily routine for eight weeks and to record their physical activities.

INTERVENTIONS:
Behavioral: Exergame Training — The individualized exergames were designed for a pressure sensitive plate connected to a personal computer and a frontal screen. The pressure-sensitive plate allows a precise analysis of the user's movements. This concurrent motor-cognitive training aims to improve motor and cognitive functions in an ecological valid setting. The cognitive functions are triggered by specific stimuli in the game scenarios. The video games are controlled via specific (whole body) movements as steps, weight shifting, jumps, and arm movements. The training focus is mainly on multi-tasking, balance and coordination as well as executive functions and attention. Furthermore, the meaningful games (colorful and appealing visuals) were designed to motivate the players to move. As the exergame will automatically adapt (individual progression) during play time, participants are challenged at their individual motor and cognitive level.
  Arms: Intervention

SUMMARY:
This study examines the feasibility and preliminary effects of user-centered exergames (video game-based physical exercise) in persons with multiple sclerosis (PwMS). The user-centered exergames were developed within a interdisciplinary team to meet the requirements of the end-users. The individualized exergames were designed for the Dividat Senso, a pressure sensitive plate connected to a personal computer and a frontal screen. This concurrent motor-cognitive training aims to improve motor and cognitive functions in an ecological valid setting. The cognitive functions are triggered by specific stimuli in the game scenarios. The video games are controlled via specific (whole body) movements as steps, weight shifting, jumps, and arm movements. The training focus is mainly on balance and coordination as well as executive functions and attention. Furthermore, the meaningful games (colorful and appealing visuals) were designed to motivate the players to move.

Participants are allocated to the either the intervention group or the control group (quasi-randomization). Participants in the intervention group perform 16 training session over a period of 4 to 8 weeks (depending on in- or out-patient). One training session lasts between 15-25 minutes. Since the difficulty of the games is adaptive to the ability level of each participant, they should neither be over- nor under-challenged. Participates in the control group continue their normal daily routine over 8 weeks. Measurements are performed before, in-between, and after the intervention period to assess feasibility parameters as well as motor and cognitive functions in all participants.

DETAILED DESCRIPTION:
The study was designed to examine the feasibility of the intervention as well as to get preliminary results about the effects of the user-centered exergame training on motor and cognitive functions in persons with multiple sclerosis (PwMS).

The entire study last 5 months (March 2021 to July 2021) and is performed in three study locations (two rehabilitation clinics and one physiotherapy).

PwMS are informed by their local physiotherapists and research associates about the study. All interested PwMS are then screened for eligibility. A sample size of 30 PwMS is anticipated where 15 participants are allocated to the intervention group and 15 participants to the control group (quasi-randomization). Measurements are performed before, in-between, and after the intervention period to assess feasibility parameters as well as motor and cognitive functions in all participants.

Intervention group:The user-centered exergames were developed within a interdisciplinary team to meet the requirements of the end-users. The individualized exergames were designed for the Dividat Senso, a pressure sensitive plate connected to a personal computer and a frontal screen. The pressure-sensitive plate allows a precise analysis of the user's movements through several high-resolution sensors. Furthermore, this plate detects position and timing information that are then used to provide the user with real-time feedback and/or game adaptations. To support users with potential balance issues and to avoid fall events, a handrail is mounted around the plate.This concurrent motor-cognitive training aims to improve motor and cognitive functions in an ecological valid setting. The cognitive functions are triggered by specific stimuli in the game scenarios. The video games are controlled via specific (whole body) movements as steps, weight shifting, jumps, and arm movements. The training focus is mainly on multi-tasking, balance and coordination as well as executive functions and attention. Furthermore, the meaningful games (colorful and appealing visuals) were designed to motivate the players to move. Participants in the intervention group perform 16 training session over a period of 4 to 8 weeks (depending on in- or out-patient). One training session lasts between 15-25 minutes. Since the difficulty of the games is adaptive to the ability level of each participant, they should neither be over- nor under-challenged. Each participant starts the exergame training at the lowest level to get familiar with the game control system. As the exergame will automatically adapt (individual progression) during play time, participants are challenged at their individual motor and cognitive level. Furthermore, participants write down the amount, type, and duration of activities besides the exergames training in an activity diary.

Control group:Participants of the control group are instructed to continue their normal daily activities over the period of eight weeks. To evaluate the amount of active time, the participants get an activity diary where they can write down the amount, type, and duration of their activities.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MS
* Able to provide written informed consent and understand instructions
* Able to play the exergames by stepping and weight shifting
* Able to walk at least 12m with or without walking aid
* Visual acuity with correction sufficient to work on a TV screen

Exclusion Criteria:

* Presence of musculoskeletal conditions that affect training performance
* Excessive fatigue that impairs training participation
* Exercise intolerance that prevents training participation
* Rapidly progressive or terminal illness
* Acute or unstable chronic illness

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-28 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessed by recruitment rate | Through recruitment completion, an average of 12 weeks
  Recruitment rate is the number of study participants compared to the number of initial planned participants
Feasibility assessed by adherence rate | Through intervention completion, 4 to 8 weeks (depending on in- and outpatient)
  Adherence rate is the number of attended training sessions compared to the number of planned trainings
Feasibility assessed by attrition rate | Through study completion, an average of 20 weeks
  Attrition rate is the number of dropouts
Feasibility assessed by a safety protocol | Through study completion, an average of 20 weeks
  Safety protocol includes number of adverse events (including serious adverse events) and specific questions about safety issues
System Usability | Through study completion, an average of 20 weeks
  The System Usability Scale interprets the system usability from 1 to 100, similar to a percentage score. A SUS score of at least 70 has to be reached to have an "acceptable" solution (52 = ok, 73 = good, 85 = excellent, 100 = best imaginable).
  The SUS consists of 10 items on a 5-point Likert scale and lasts about 3 minutes.
  The SUS is assessed at post-measurement.
Feasibility, usability and training experience - Semi-structured interview | Through study completion, an average of 20 weeks
  The semi-structured interview contains pre-defined questions about user's gameplay experiences related to their body, controller, experience, virtual game scenario and safety.
  The interview lasts about 20 minutes and is assessed at post-measurement.

SECONDARY OUTCOMES:
Changes in balance and mobility | Through study completion, an average of 20 weeks
  Balance and mobility are assessed with the Timed Up and Go Test. Time needed to complete the assessment is recorded.
  Test duration is about 5 to 10 minutes and is assessed at pre- and post-measurement.
Changes in spatio-temporal gait parameters | Through study completion, an average of 20 weeks
  Gait analysis is conducted under single (walking; normal speed) and dual (walking + counting; normal speed) over 13 meters to assess spatio-temproal gait parameters ((gait speed, step length, gait variability and double support time).
  Gait parameters are assessed via the system Physiolog. Test duration is about 10 to 15 minutes and is assessed at pre- and post-measurement.
Changes in information processing speed | Through study completion, an average of 20 weeks
  Simple reaction time test is performed on a personal computer recording reaction time [ms] and errors.
  Test duration is about 5 minutes and is assessed at pre- and post-measurement.
Changes in executive functions - inhibition | Through study completion, an average of 20 weeks
  Flanker test is performed on a personal computer recording reaction time [ms] and errors.
  Test duration is about 10 minutes and is assessed at pre- and post-measurement.
Changes in executive functions - flexibility | Through study completion, an average of 20 weeks
  Trail Making Test A & B is performed on a personal computer recording reaction time [ms] and errors.
  Test duration is about 10 minutes and is assessed at pre- and post-measurement.
Training experience - Physical Activity Enjoyment Scale | Through study completion, an average of 20 weeks
  The Physical Activity Enjoyment Scale (PACES) measures enjoyment in physical activity environments.
  The PACES consists of 18 bipolar items on a 7-point Likert scale, lasts about 5 minutes, and is assessed after the first and last training session
Training experience - Flow Short Scale | Through study completion, an average of 20 weeks
  The Flow Short Scale (FFS) assesses the flow experience for training experiences.
  The FSS consists of 13 items on a 5-point Likert scale and lasts about 5 minutes, and is assessed after the first and last training session.

OTHER OUTCOMES:
Training parameters | Through intervention completion, 4 to 8 weeks (depending on in- and outpatient)
  Training parameters such as level, points, play time per session, type of game and dual task or single task are collected in a training protocol.
  The use (always, sometime or not) of the handrail is noted.
Training intensity | Through intervention completion, 4 to 8 weeks (depending on in- and outpatient)
  Training intensity is rated on a 10-point rating scale (1 = very weak, 10 = very,very strong) to assess the perceived cognitive and physical exertion.
Training progress | Through intervention completion, 4 to 8 weeks (depending on in- and outpatient)
  The training progress is assessed by video recordings. With these video recordings possible deficiencies or difficulties can be detected.
Demographic and medical data | Through study completion, an average of 20 weeks
  The questionnaire assesses general personal information about participants covering general health, medical history and physical activity.
  The survey lasts about 10 minutes and is assessed at pre-measurement.
Activities-specific Balance Confidence | Through study completion, an average of 20 weeks
  Activities-specific Balance Confidence (ABC) scale assesses the confidence in doing different activities without losing the balance or becoming unsteady.
  The ABC scale consists of 16 items where each item is rated from 0% (not confident) to 100% (very confident) and lasts about 5 minutes and is assessed at pre-measurement.
Multiple Sclerosis Impact | Through study completion, an average of 20 weeks
  The Multiple Sclerosis Impact Scale (MSIS) assesses the physical and psychological impact of MS.
  The MSIS consists of 29 items on a 5-point Likert scale, lasts about 10 minutes and is assessed at pre-measurement.
Fatigue | Through study completion, an average of 20 weeks
  The Fatigue Severity Scale (FSSc) assesses the degree of fatigue. The FSSc consists of 9 items on a 7-point Likert scale, lasts about 3 minutes and is assessed at pre-measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zürich, Zurich, Switzerland